CLINICAL TRIAL: NCT07130929
Title: Intensive Rehabilitation by Functional Electrical Stimulation for the Treatment of Critical Neuromyopathy in Patients With Severe Stroke Admitted to the Highly Specialized Intensive Rehabilitation Unit: a Pilot Study
Brief Title: Functional Electrical Stimulation to Treat Critical Neuromyopathy After Severe Stroke: a Pilot Study.
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RISE
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Intensive Care Unit (ICU) Acquired Weakness (ICU - AW); Acquired Brain Injury (Including Stroke)
Keywords: stroke; Intensive Care Unit (ICU) acquired weakness (ICU - AW); Functional Electrical Stimulation; FES; Rehabilitation
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm in treatment with conventional physiotherapy plus FES (Experimental)
  Interventions: Other: Functional Electrical Stimulation
- Arm in treatment with only conventional physiotherapy (Active Comparator): conventional physiotherapy in an equivalent additional session (without FES).
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Functional Electrical Stimulation — Physiotherapy exercises, selected from a group of active flexion-extension exercises, cycle ergometer, sit-to-stand exercises and a preparatory exercise for the gait pattern with hip flexion and subsequent loading on the lower limb, associated with functional electrical stimulation.
  Arms: Arm in treatment with conventional physiotherapy plus FES
Other: Conventional physiotherapy — Conventional physiotherapy exercises, selected from a group of active flexion-extension exercises, cycle ergometer, sit-to-stand exercises and a preparatory exercise for the gait pattern with hip flexion and subsequent loading on the lower limb.
  Arms: Arm in treatment with only conventional physiotherapy

SUMMARY:
This study aims to evaluate the effectiveness of physiotherapy treatment combined with functional electrical stimulation (FES) in a small group of patients with severe acquired brain injury (SABI) of vascular origin and with a clinical and instrumental diagnosis of "Intensive Care Unit-Acquired Weakness" (ICU-AW). Functional electrical stimulation is a technology that uses electrical impulses, generated by an external device, to reactivate the neuromuscular system through electrodes applied to the skin. In functional electrical stimulation, this process is integrated into physiotherapy sessions, with the active involvement of the patient, through the performance of exercises with the assistance and supervision of the physiotherapist. The rationale behind this is to stimulate neuroplasticity processes by facilitating movement through the application of electrical stimuli and the active participation of the patient in performing a motor task, in an attempt to promote improvement in an impaired function.

In particular, the objectives that will be pursued are: improvement of lower limb neuromyopathy assessed clinically using the Medical Research Council (MRC) scale, the Fugl-Meyer scale for lower limbs, the Short Physical Performance Battery (SPPB) scale, the assessment of active and passive Range Of Motion (ROM) of the main joints of the lower limb (hip, knee, ankle) and measured instrumentally by neurophysiological examination and ultrasound examination.

After randomization, patients in the control arm will be treated with physiotherapy and speech therapy sessions as per the conventional protocol, and an additional 15 physiotherapy sessions lasting 60 minutes over a period of 5 weeks. Alternatively, patients in the experimental group will receive, in addition to conventional rehabilitation treatment, a treatment consisting of 15 physiotherapy sessions combined with FES lasting 60 minutes over a period of 5 weeks.

At the end of the treatment period, baseline characteristics and clinical and instrumental outcome variables will be compared between the two groups using the chi-square test for dichotomous and categorical variables and the t-test for independent samples or the Mann-Whitney U test for continuous variables, depending on whether or not they are normally distributed. In all analyses, a p-value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic vascular GCA involving unilateral motor deficit < 3 months;
* Premorbid Modified Rankin Scale <2;
* Age >18 years and <80 years;
* Level of Cognitive Functioning > 4 for active participation in treatment.
* MRC total sum score <= 48 (range 0 -60) for clinical suspicion of ICU-AW
* Clinical diagnosis of tetra/paraparesis of peripheral origin confirmed by neurophysiological examination;
* Signature of informed consent by the patient or, if incapacitated, by their legal representative.

Exclusion Criteria:

* Clinical cardio-respiratory or internal instability such as to prevent treatment;
* History of previous comorbidity for ICU-AW;
* Previous known chronic neuropathy;
* Severe coagulopathy;
* Skin integrity problems at the interface surfaces with the electrostimulator;
* Epilepsy not controlled by medication;
* Presence of implanted electronic devices;
* Pregnancy or breastfeeding;
* Severe spasticity with a score of >3 on the modified Ashworth scale;
* Treatment with botulinum toxin;
* Recent malignant neoplasm;
* Conditions that put you at risk for neuropathies, e.g., history of diabetes mellitus, renal failure, hepatic failure, vitamin deficiencies, chronic alcoholism, vasculitis, previous use of neurotoxic drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Change in lower limb neuromyopathy assessed blindly compared to the treatment/control arm at the clinical level using the Medical Research Council (MRC) scale. | From enrollment to the end of treatment at 5 weeks from T0 (T1) and from enrollment to the follow-up at 12 weeks from T0(T2).

SECONDARY OUTCOMES:
Change in the units of the scale "Fugl-Meyer scale for lower limbs". | From enrollment to the end of treatment at 5 weeks (T1) and from enrollment to the follow-up at 12 weeks(T2).
Change in the units of the scale "the Short Physical Performance Battery (SPPB) scale". | From enrollment to the end of treatment at 5 weeks from T0 (T1) and from enrollment to the follow-up at 12 weeks from T0(T2).
Change in the degrees of the active range of motion of the main joints of the lower limbs (hip, knee, ankle). | From enrollment to the end of treatment at 5 weeks from T0 (T1) and from enrollment to the follow-up at 12 weeks from T0(T2).
Change in the degrees of passive range of motion of the main joints of the lower limbs (hip, knee, ankle). | From enrollment to the end of treatment at 5 weeks from T0 (T1) and from enrollment to the follow-up at 12 weeks from T0(T2).
Change in the parameters recorded during the neurophysiological examination using electromyography. | From enrollment to the end of treatment at 5 weeks (T1).
Change in the parameters recorded during ultrasound examination | From enrollment to the end of treatment at 5 weeks (T1).
  Change in the parameters recorded during ultrasound examination of the transverse diameter of the rectus femoris.
Change in the parameters recorded during ultrasound examination | From enrollment to the end of treatment at 5 weeks
  Change in the difference between the distance from the skin plane and the deep layer of the rectus femoris recorded with the muscle at rest and during contraction, recorded using M-mode ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS-Fondazione Don Gnocchi, Florence, FI, Italy

REFERENCES:
- [Background] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139
- [Background] Cecatto RB, Maximino JR, Chadi G. Motor recovery and cortical plasticity after functional electrical stimulation in a rat model of focal stroke. Am J Phys Med Rehabil. 2014 Sep;93(9):791-800. doi: 10.1097/PHM.0000000000000104. PMID 24800715
- [Background] Peckham PH, Knutson JS. Functional electrical stimulation for neuromuscular applications. Annu Rev Biomed Eng. 2005;7:327-60. doi: 10.1146/annurev.bioeng.6.040803.140103. PMID 16004574
- [Background] Intiso D, DI Rienzo F, Fontana A, Tolfa M, Bartolo M, Copetti M. Functional outcome of critical illness polyneuropathy in patients affected by severe brain injury. Eur J Phys Rehabil Med. 2017 Dec;53(6):910-919. doi: 10.23736/S1973-9087.17.04595-6. Epub 2017 Apr 14. PMID 28417610
- [Background] Hakiki B, Draghi F, Scarpino M, Portaccio E, Romoli A, Mannini A, Atzori T, Lolli F, Macchi C, Grippo A. Critical illness polyneuromyopathy: Functional impact after severe acquired brain injuries. Acta Neurol Scand. 2020 Dec;142(6):574-584. doi: 10.1111/ane.13324. Epub 2020 Aug 31. PMID 32740902